CLINICAL TRIAL: NCT02555631
Title: Translating the Diabetes Prevention Program to Engage Men From Disadvantaged Areas
Brief Title: PowerUp for Health: A Diabetes Prevention Program for Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: The New York Academy of Medicine (Other); University of Pittsburgh (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Elizabeth Walker, Professor of Medicine, Albert Einstein College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2014-3604; R18DK102080 (NIH)
Record Dates: First submitted 2015-09-17; First posted 2015-09-21 (Estimated); Results first posted 2018-06-28 (Actual); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: Type 2 Diabetes; Men
Keywords: type 2 diabetes; prevention; men
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Multiple Endocrine Neoplasia Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- lifestyle intervention (Experimental): In this pilot study, each subject will receive the lifestyle intervention of the diabetes prevention program, a modified program for men from disadvantaged neighborhoods--a 16 weekly sessions of 1 hour each session
  Interventions: Behavioral: lifestyle

INTERVENTIONS:
Behavioral: lifestyle — In this pilot study, each subject will receive the lifestyle intervention of the diabetes prevention program, a modified program for men from disadvantaged neighborhoods--a 16 weekly sessions of 1 hour each session

SUMMARY:
The purpose of this two-year proposal is to:

1. develop and
2. complete a pilot test of an adaptation of the evidence-based National Diabetes Prevention Program (NDPP) tailored to engage men with prediabetes in disadvantaged communities in New York City.

The sites for this pilot study are New York City Parks and recreation centers. Study's main outcome is weight loss of 5-7% baseline weight.

DETAILED DESCRIPTION:
During year one, the multi-disciplinary research team will work closely with the expert and community Advisory Panel and consultants to adapt the standard NDPP curriculum in order to promote increased engagement of men. "Engagement" is defined in this proposal to include recruitment, group participation and retention in the 16-week program. This modified NDPP♂ (i.e., for men) renamed by the advisory panel as "Power Up for Health," will have only NDPP-trained male coaches and male participants, with adaptations to dietary and physical activity messaging and a new behavioral "toolbox" approach developed for men.

By month 10 of year one, investigators will begin implementation of the 16-week pilot studies of the NDPP♂ at 6 NYC Parks and Recreation Department (REC) sites in disadvantaged communities in three of the NYC boroughs currently offering the standard NDPP programming. Investigators will utilize an iterative and adaptive process during the pilot phase to modify recruitment and retention strategies, as well as the NDPP curriculum and activities. The exploratory aim, as feasible, is to then compare the adapted NDPP♂ pilot data to the standard NDPP mixed-gender groups' available data on recruitment, participation, weight loss, and retention of men from similar NYC neighborhoods. The goal will be pilot study data from 15-20 male participants at each REC pilot site-a recruitment goal of 120 male participants. Working in collaboration with the investigators' consultants and Advisory Panel of community leaders and academic experts in men's health promotion, as well as study partners at the NYC Department of Parks and Recreation, investigators will conduct focused outreach to the target populations.

The Specific Aims for the Pilot Study are:

Aim 1. to collaborate with the expert and community Advisory Panel to complete the adaptation of the NDPP curriculum and the recruitment and retention activities to better engage men with prediabetes from disadvantaged communities of NYC;

Aim 2. to assess preliminary indicators of effectiveness of the NDPP♂ with respect to reductions in body weight; Hypothesis 1: Men engaged in the NDPP♂ will have reductions in body weight at 16 weeks at least equivalent to the NDPP goal of 5-7% of their baseline body weight.

Aim 3. to examine and describe from pilot data the extent to which recruitment, intervention and retention strategies, tailored for men with prediabetes are associated with improved engagement of the target population; Exploratory Hypothesis 3.1: Recruitment of men to NDPP♂ will occur more rapidly and with less intensive strategies than recruitment of men to the standard NDPP in comparable communities.

Exploratory Hypothesis 3.2: Men enrolled in the NDPP♂ will be more engaged in program activities and self-report greater improvements in healthy eating and physical activity compared with men in the standard NDPP.

Exploratory Hypothesis 3.3: Men enrolled in the NDPP♂ will have retention rates that are at least equivalent to men in the standard NDPP.

All comparison data analyses are exploratory and as data are available.

Aim 4. to examine preliminary data to identify demographic, psychosocial, neighborhood, and REC site characteristics associated with differential recruitment, retention and intervention effects in the NDPP♂.

ELIGIBILITY:
Inclusion Criteria:

* pre-diabetes by ADA risk test or an A1c in past year in prediabetes range
* BMI 24 or above (22 for Asians)
* male
* lives, works or spend much time in the disadvantaged neighborhood of the park site

Exclusion Criteria:

* cannot read or write in English or Spanish
* has diagnosed diabetes
* obvious mental disability so as to preclude health behavior changes

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2015-09; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A. Walker, PhD, RN, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein College of Medicine, The Bronx, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lifestyle Intervention
Started | 29
Completed | 25
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Lifestyle Intervention
Number analyzed (Participants) | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.9 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 29
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Change in Weight in Pounds
Description: the goal is to lose 5-7% of baseline body weight for pre-diabetic men
Time Frame: Baseline, 16 weeks
Measure: Mean (Full Range); unit: percentage of body weight lost
Arm/Group | Lifestyle Intervention
Number analyzed (Participants) | 25
percentage of body weight lost | 3.8 [-0.2 to 8.1]

2. Secondary Outcome: Number of Men Enrolled During 8 Weeks of Recruitment
Description: measured by numbers of men and the timeframe in which the recruitment takes place;
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Lifestyle Intervention
Number analyzed (Participants) | 29
Participants | 29

3. Secondary Outcome: Number of Sessions Attended
Description: with a measured goal of at least attendance observed and recorded at 9/16 sessions on average
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: Sessions Attended
Arm/Group | Lifestyle Intervention
Number analyzed (Participants) | 25
Sessions Attended | 11.7 (3.9)

4. Secondary Outcome: Number of Participants That Participated in Each Session
Description: this is measured by direct observation at selected sessions; report by the lifestyle coach; and discussion during focus groups at the end of the 16 weeks
Time Frame: 16 weeks
Measure: Number; unit: Participants
Arm/Group | Lifestyle Intervention
Number analyzed (Participants) | 25
Participants | 25

ADVERSE EVENTS:
Arm/Group | Lifestyle Intervention
Serious Adverse Events (participants affected / at risk) | 0/29
Other Adverse Events (participants affected / at risk) | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes